CLINICAL TRIAL: NCT01042158
Title: A Clinical Trial of Ambrisentan and Tadalafil in Pulmonary Arterial Hypertension Associated With Systemic Sclerosis
Acronym: ATPAHSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eli Lilly and Company (Industry); United Therapeutics (Industry); The Cleveland Clinic (Other); University of Texas (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAD-PH-001; P50HL084946 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Arterial Hypertension; Systemic Sclerosis; Scleroderma Spectrum of Diseases; Connective Tissue Disease; Pulmonary Hypertension
Keywords: Tadalafil; Ambrisentan; Quality of Life
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Scleroderma, Systemic; Connective Tissue Diseases; Hypertension, Pulmonary | interventions — Tadalafil; ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tadalafil and ambrisentan upfront therapy (Other): This will be a 36-week, single group, open label study assessing the effects of Tadalafil plus Ambrisentan combination therapy in patients with pulmonary arterial hypertension associated with the scleroderma spectrum of disease (PAH-SSD).
  Interventions: Drug: tadalafil and ambrisentan upfront combination therapy

INTERVENTIONS:
Drug: tadalafil and ambrisentan upfront combination therapy — tadalafil 20 mg qd and ambrisentan 5 mg qd. Up-titration of study medications will occur at week 4 (ambrisentan 10 mgs daily and tadalafil 40 mg qd). If a subject experiences an intolerable adverse event as a result of an uptitration in the study drug dose, the dose of study drug maybe down titrated to 20 mg of tadalafil and/or 5mg of ambrisentan. If the subject is still experiencing an intolerable adverse event, then the investigator will withdraw the subject from the study.
  Other Names: Adcirca; Letairis

SUMMARY:
This will be a 36-week, single group, open label study assessing the effects of Tadalafil plus Ambrisentan combination therapy in patients with pulmonary arterial hypertension associated with the scleroderma spectrum of disease (PAH-SSD). Standard outcome measures such as six-minute walk distance (6MWD), New York heart Association (NYHA) classification, and hemodynamic measurements will be assessed, as well as novel functional measures of RV-PV function including the transthoracic echocardiogram parameter tricuspid annular plane systolic ejection (TAPSE), contrast-enhanced cardiac MRI and heart rate variability assessed by Holter monitoring. This design (excluding a placebo arm) was selected for ethical concerns and to provide optimal efficiency and active therapy to all study subjects. It also allows for comparisons between the two monotherapies and with combination therapy.

DETAILED DESCRIPTION:
Pulmonary Arterial Hypertension (PAH) includes a heterogeneous group of clinical entities sharing similar clinical and pathological features that have been subcategorized as idiopathic PAH (IPAH, formerly known as "primary pulmonary hypertension" or PPH), familial PAH, pulmonary hypertension related to connective tissue diseases (such as systemic sclerosis), portopulmonary hypertension and pulmonary hypertension related to HIV infection, drugs and toxins (10). PAH is clinically defined by a resting mean pulmonary artery pressure ≥ 25 mmHg and pulmonary artery wedge pressure ≤ 15 mmHg in the absence of left heart disease, underlying parenchymal lung disease, thromboembolic disease or other causes of pulmonary hypertension.

PAH is characterized by increased pulmonary vascular resistance due to remodeling and occlusion of the pulmonary arterioles. Left untreated, PAH leads irremediably to right ventricular (RV) hypertrophy, pressure overload and dilation resulting in death within 2-3 years (11). For the past two decades, it has been appreciated that the integrity of the RV function, rather than the degree of pulmonary vascular injury, is the major determinant of symptoms and mortality in patients with PAH. RV dysfunction at time of presentation, as reflected by an elevation in right atrial pressure (RAP), the presence of pericardial effusion or depressed cardiac output (CO), is a powerful prognosticator of death (12).

Current PAH therapies consist of prostacyclin analogues, endothelin receptor antagonists (ETRA) and phosphodiesterase type V (PDE V) inhibitors (13). All have been shown to be effective in improving exercise capacity as measured by the 6 MWD in short term (12 - 16 week) randomized, placebo-controlled clinical trials. However, the clinical response is highly variable and mortality remains high (14). Moreover, the majority of subjects enrolled in these trials have had IPAH. Over the past 10 years, the Johns Hopkins Pulmonary Hypertension Program and Scleroderma Center have worked closely to address the daunting clinical challenge of PAH associated with scleroderma or systemic sclerosis (PAH-SSc). Previous work from our group (15;16) and others (17-19) has clearly demonstrated a markedly worse prognosis in PAH-SSc compared with IPAH despite similar treatments. An intriguing and consistent finding when comparing these two groups is that whereas mPAP is, on average, lower in PAH-SSc, markers of RV dysfunction (e.g. CO and RAP) are similar, raising the possibility of maladaptive RV response to pressure overload and/or intrinsic myocardial disease. Current PAH therapies target pathways that have been implicated in the remodeling of the pulmonary vasculature (PV). However, there is no clear evidence that these therapies have altered PV and/or RV remodeling or offered significant beneficial effects in patients with PAH-SSc in whom mortality remains exceedingly high. In addition, their effects on RV dysfunction and RV-PV interaction remain poorly characterized.

We hypothesize that improvement in PAH-SSc will only be achieved with therapy directly targeted at RV-PV dysfunction. Sildenafil and tadalafil inhibit phosphodiesterase type 5 (PDE5) which is abundant in the lung and is the main enzyme responsible for cyclic Guanosine MonoPhosphate (cGMP) hydrolysis. The resulting increase in cGMP probably mediates the relaxant and anti-hypertrophic actions of nitric oxide and natriuretic peptides in vascular tissues, and exerts a direct anti-hypertrophic action on cardiac muscle as demonstrated in compelling preliminary experiments by investigators of the NHLBI-funded Hopkins Scientific Center of Clinically Oriented Research (SCCOR) in Pulmonary Vascular Disease. In these experiments, sildenafil was capable of preventing and reversing RV hypertrophy and dysfunction in a model of pulmonary artery banding, similar to its effects on the left ventricle with aortic banding (20), indicating a direct beneficial action on RV remodeling.

Both sildenafil (21) and tadalafil (22) have been demonstrated to be effective in PAH and are FDA approved for this indication. The endothelin-receptor antagonists, bosentan (23) and ambrisentan (24), are also FDA-labeled for this indication and represent alternative options for oral therapy of PAH (25). A small randomized study comparing sildenafil with bosentan suggested that sildenafil was superior in reducing RV mass and improving exercise capacity in patients with PAH (26). Recently, the results of a large multi-center randomized, controlled trial of tadalafil therapy for PAH have been presented. The data indicate, that similar to sildenafil, tadalafil at doses of 20 and 40 mg per day, improved exercise capacity. In addition, tadalafil 40 mg per day improved pulmonary hemodynamics, quality of life and reduced the incidence of clinical worsening.

This study aims to compare the effects of upfront combination therapy with tadalafil and ambrisentan in PAH-SSc on PVR and RV mass. It will also assess novel markers of RV function by cardiac MRI and echocardiography, as well as the conventional endpoints, including 6 MWD and functional class. The trial is unique in that it will enroll only PAH-SSc patients, the PAH subgroup with the poorest outcomes and will be considerably longer in duration (36 weeks) than previous studies.

ELIGIBILITY:
Inclusion Criteria:

* A right heart catheterization done at baseline with a mean pulmonary artery pressure (mPAP) ≥ 25mmHg, pulmonary artery wedge pressure (PAWP) ≤ 15mmHg, and pulmonary vascular resistance (PVR) ≥3 Woods units.
* Scleroderma defined as systemic sclerosis with diffuse or limited scleroderma meeting the American College of Rheumatology (ACR) criteria (33). Cases will be included if they meet clinical features that satisfy ACR criteria for a diagnosis of scleroderma or the presence of three of five features of the CREST syndrome are identified; or there is the presence of definite Raynaud's phenomenon, abnormal nail fold capillaries typical of scleroderma and the presence of a specific scleroderma related auto-antibody. Limited skin involvement is defined as skin tightening distal to elbows and knees with or without facial involvement; and diffuse skin involvement, tightening proximal to these joints or truncal involvement.
* Subjects will be older than 18 years of age with a diagnosis of PAH-SSc.
* Subjects will be NYHA functional class II or III.
* 6 minute walk distance ≥ 100 meters and ≤ 500 meters at screening and baseline.
* Negative urine pregnancy test for women of childbearing age at screening and baseline visits.
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Right heart catheterization reveals evidence of pulmonary venous hypertension (pulmonary capillary wedge pressure > 15 mm Hg).
* Significant chronic obstructive: Forced expiratory volume in 1 second to forced expiratory volume ratio < 70% and a forced expiratory volume in 1 second less than 60% of predicted.
* Interstitial lung disease

  1. Based on a combination of pulmonary function tests and chest radiography.
  2. Patients will be excluded if they have a total lung capacity less than 60% of predicted and included if the total lung capacity was ≥ 70%. Patients with a total lung capacity between 60 and 70% of predicted are included if their computed tomography scan demonstrates only minimal interstitial fibrosis
* Portal hypertension.
* Severe obstructive sleep apnea.
* Chronic thromboembolic disease.
* Positive antibodies to the human immunodeficiency virus.
* History of anorexigen use including fen-phen.
* Any other disease known to be associated with pulmonary hypertension.
* Subjects with other etiology for pulmonary hypertension besides PAH-SSc.
* Subjects with liver function abnormalities (ALT or Aspartate Aminotransferase (AST) > 3 times the upper limit of normal at screening or at baseline) or chronic liver disease.
* Advanced kidney failure (GFR < 30 ml/min at screening or at baseline).
* Acute decompensation of underlying illness or hospitalization for pulmonary hypertension within 4 weeks prior to enrollment.
* Prior chronic therapy with an endothelin-receptor antagonist, PDE V inhibitor, or a prostacyclin analogue.
* History of hypersensitivity reaction or adverse effect related to ambrisentan or tadalafil.
* History of implantable permanent pacemaker or any metallic objects in the body.
* Participation in a clinical study involving an investigational drug or device within four weeks before the screening visit.
* Pregnant or lactating women.
* Concomitant use of nitrates (any form) either regularly or intermittently
* Concomitant use of potent Cytochrome P3A (CYP3A) inhibitors (eg, ritonavir, ketoconazole, itraconazole)
* Any additional contraindications and precautions specified in the package inserts for Tadalafil (Adcirca) and Ambrisentan (Letairis) not listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hassoun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sato T, Ambale-Venkatesh B, Lima JAC, Zimmerman SL, Tedford RJ, Fujii T, Hulme OL, Pullins EH, Corona-Villalobos CP, Zamanian RT, Minai OA, Girgis RE, Chin K, Khair R, Damico RL, Kolb TM, Mathai SC, Hassoun PM. The impact of ambrisentan and tadalafil upfront combination therapy on cardiac function in scleroderma associated pulmonary arterial hypertension patients: cardiac magnetic resonance feature tracking study. Pulm Circ. 2018 Jan-Mar;8(1):2045893217748307. doi: 10.1177/2045893217748307. Epub 2017 Dec 18. PMID 29251556
- [Derived] Hassoun PM, Zamanian RT, Damico R, Lechtzin N, Khair R, Kolb TM, Tedford RJ, Hulme OL, Housten T, Pisanello C, Sato T, Pullins EH, Corona-Villalobos CP, Zimmerman SL, Gashouta MA, Minai OA, Torres F, Girgis RE, Chin K, Mathai SC. Ambrisentan and Tadalafil Up-front Combination Therapy in Scleroderma-associated Pulmonary Arterial Hypertension. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1102-10. doi: 10.1164/rccm.201507-1398OC. PMID 26360334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had recruitment of patients from four centers, namely Johns Hopkins University, Stanford University, University of Texas Southwestern Medical Center, and the Cleveland Clinic. Patients who fulfilled the inclusion and exclusion criteria were screened for enrollment between August 25, 2011 and February 4, 2014.
Pre-assignment Details: This was a one arm study and patients were therefore selected based on the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Started | 25
Completed | 24
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Right Ventricular (RV) Mass
Description: Assessment of change in Right ventricular mass was done via standard volumetric cine images of the right heart at baseline and comparing it to that at the end of 36 weeks using Cardiac Magnetic Resonance Imaging studies.
Time Frame: baseline and 36 weeks
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Number analyzed (Participants) | 24
grams
  Baseline | 32.5 [23.2 to 41.4]
  At 36 weeks | 28.0 [20.6 to 32.9]

2. Primary Outcome: Pulmonary Vascular Resistance (PVR)
Description: Change in Pulmonary Vascular Resistance (PVR) was ascertained via Right Heart Catheterization (RHC) measurement of the difference between the PVR at baseline and 36 weeks
Time Frame: baseline 36 weeks
Measure: Median (Inter-Quartile Range); unit: Wood units
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Number analyzed (Participants) | 24
Wood units
  Baseline | 6.9 [4.0 to 12.9]
  At 36 weeks | 3.1 [2.0 to 5.7]

3. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE)
Description: The extent of displacement of the tricuspid valves, termed as Tricuspid Annular Plane Systolic Excursion (TAPSE) was measured using a trans-thoracic echocardiogram following Right heart catheterization.
Time Frame: baseline and 36 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Number analyzed (Participants) | 24
cm
  Baseline at week 0 | 2.2 (0.12)
  week 36 | 1.65 (0.11)

4. Secondary Outcome: 6-minute Walk Distance
Description: patients were made to take a walk of normal speed to cover a distance in 6 minutes and distance covered was recorded. This was done at baseline (week o) and then repeated t 36 weeks.
Time Frame: baseline and 36 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
Number analyzed (Participants) | 24
meters
  Baseline (week 0) | 343 (131)
  Week 36 | 395 (99)

ADVERSE EVENTS:
Time Frame: through study completion, up to 36 weeks
Arm/Group | Tadalafil and Ambrisentan Upfront Therapy
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil and Ambrisentan Upfront Therapy (N=24)
Stenosis of the left internal carotid artery, worsening shortness of breath, Right heart failure (Cardiac disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
1. An open-label study with no placebo group
2. Relatively small number of patients and therefore vulnerable to confounding natural history with treatment effects
3. Measurements performed at four different institutions
4. Few missing data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No